CLINICAL TRIAL: NCT02246907
Title: Effects of Exercise on Patient Reported Outcomes in Newly Diagnosed Adults With Acute Leukemia During Induction Treatment: Exercise and Quality of Life in Leukemia Patients (EQUAL)
Brief Title: Exercise and Quality of Life in Leukemia Patients
Acronym: EQUAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC1234
Record Dates: First submitted 2014-03-27; First posted 2014-09-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Acute Leukemia
Keywords: Health related quality of life
MeSH Terms: interventions — Exercise; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): The control group will receive standard of care which includes recreational therapy and standard encouragement.
- Exercise (Other): Participants in this arm will receive standard of care plus exercise for the duration of their inpatient stay for induction chemotherapy.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — All intervention patients will participate in an individualized prescriptive exercise intervention 2 to 4 times per week for a period of the induction chemotherapy/in-hospital recovery. The exercise intervention will begin on week 1 of the study, the day after the first batteries of initial assessments are concluded. Each exercise session will be divided into two parts. One part will be administered in the morning and the second one late in the afternoon. There will be a period of rest of at least 36 hours between each exercise session.
  Other Names: Exercise and Quality of Life in Acute Leukemia Patients
  Arms: Exercise

SUMMARY:
The purpose of this study is to evaluate the impact of an exercise intervention on patient-reported anxiety, depression, fatigue, and sleep disturbances among acute leukemia patients. The investigators hypothesize that exercise will reduce fatigue in acute leukemia patients.

DETAILED DESCRIPTION:
The purpose of this randomized, prospective, longitudinal study is to evaluate the impact of an exercise intervention on patient-reported anxiety, depression, fatigue, and sleep disturbances outcomes among acute leukemia patients. The study will include 2 groups for a total sample size of 30: n=15 control group and n=15 intervention group. Each patient enrolled in the intervention arm will participate in an exercise program for the duration of their hospitalization, 4-6 weeks on average during the first treatment (induction chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with acute leukemia by pathology report
* Admitted for induction chemotherapy within in the previous 96 hours or +/- 3 days from initiation of induction chemotherapy
* An expected hospital stay of 3-4 weeks or longer
* Participation in the study must be approved by the physician directly responsible for the patient's care while at University of North Carolina -Hospitals
* Age >21 years of age
* Willing and able to provide, signed informed consent
* Willing and able to use a computer to complete study questionnaires
* Ability to understand and speak English

Exclusion Criteria:

The criteria below will be determined by the patient's physician and a review of the patient's medical history. If any of the exclusion criteria are observed, the patients will be informed and excluded from participating in the study.

Participation in this study will involve the same risks as any exercise regimen. Given the potential risks involved, patients will be screened for exclusion based upon the following criteria:

* Cardiovascular disease (unless the disease would not compromise the patient's ability to participate in the exercise rehabilitation program)
* Acute or chronic respiratory disease that would compromise the patient's ability to participate in the exercise rehabilitation program
* Acute or chronic bone, joint, or muscular abnormalities that would compromise the patient's ability to participate in the exercise rehabilitation program
* Inability to understand and speak English
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Another active malignancy
* Patients will also be excluded if they have active bleeding, acute thrombosis, ischemia, hemodynamically unstable, and uncontrolled pain.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Compare symptoms of fatigue in newly diagnosed acute leukemia patients | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Symptoms will be assessed by patient reported survey at baseline, weekly through patient hospitalization, and then again at patient's first appointment after hospital discharge. We are interested in how the symptom changes over time.

SECONDARY OUTCOMES:
Evaluate health-related quality of life changes over time | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Health related quality of life will be assessed by patient reported survey at baseline, and at the week 4 timepoint. We are interested in change over time between groups
Compare symptoms of anxiety between groups | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Symptoms will be assessed by patient reported survey at baseline, weekly during hospitalization, and at first clinic visit after discharge from hospital. We are interested in change over time between groups.
Compare symptoms of depression between groups | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Symptoms will be assessed by patient reported survey at baseline, weekly during hospitalization, and at first clinic visit after discharge from hospital. We are interested in change over time between groups.
Compare sleep quality between groups | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Symptoms will be assessed by patient reported survey at baseline, weekly during hospitalization, and at first clinic visit after discharge from hospital. We are interested in change over time between groups.
Changes in cardiovascular function | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Exercise testing which will assess the outcome measures will be performed at baseline, and after 4 weeks of training (for the intervention group), or at the week 4 time point (for the control group). We are interested in change over time between groups.
Changes in muscle strength | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Exercise testing which will assess the outcome measures will be performed at baseline, and after 4 weeks of training (for the intervention group), or at the week 4 time point (for the control group). We are interested in change over time between groups.
Changes in body composition | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Exercise testing which will assess the outcome measures will be performed at baseline, and after 4 weeks of training (for the intervention group), or at the week 4 time point (for the control group). We are interested in change over time between groups.
Changes in functional mobility | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Exercise testing which will assess the outcome measures will be performed at baseline, and after 4 weeks of training (for the intervention group), or at the week 4 time point (for the control group). We are interested in change over time between groups.
Changes in muscle size | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Exercise testing which will assess the outcome measures will be performed at baseline, and after 4 weeks of training (for the intervention group), or at the week 4 time point (for the control group). We are interested in change over time between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Bryant, PhD, RN, Principal Investigator — UNC- Chapel Hill; Claudio Battaglini, PhD, Principal Investigator — UNC- Chapel Hill
Locations (1):
- University of North Carolina Lineberger Comprehenisive Cancer Center, Chapel Hill, North Carolina, United States